CLINICAL TRIAL: NCT04867928
Title: A Multicentric Phase 2 Study of Venetoclax and Azacitidine for the Management of Molecular Relapse/Progression in Adult NPM1-MUTATED Acute Myeloid Leukemia
Brief Title: Venetoclax and Azacitidine for the Management of Molecular Relapse/Progression in Adult NPM1-mutated Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML2521
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse; NPM1 Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax+azacitidine (Experimental): subjects will receive treatment until alloSCT
  Interventions: Drug: Venetoclax+azacitidine

INTERVENTIONS:
Drug: Venetoclax+azacitidine — subjects will receive venetoclax 400 mg orally QD on Days 1 - 28 plus azacitidine 75 mg/m2 SC or IV daily for 7 days. Cycle Length - 28 Days. . Subjects will continue treatment until subsequent alloSCT.

SUMMARY:
This is a phase 2, non-randomized, interventional, open-label, multicenter trial evaluating the efficacy of VEN-AZA as a bridge-to-transplant therapy in chemotherapy-treated adult NPM1mut AML patients who experience molecular relapse or progression during treatment or follow-up. Subjects will receive cycles of venetoclax plus azacitidine. After each cycle, MRD will be evaluated and at any time of MRD-negativity, AlloSCT will be performed.

DETAILED DESCRIPTION:
This is a phase 2, non-randomized, interventional, open-label, multicenter trial evaluating the efficacy of VEN-AZA as a bridge-to-transplant therapy in chemotherapy-treated adult NPM1mut AML patients who experience molecular relapse or progression during treatment or follow-up.

Subjects will receive venetoclax 400 mg orally QD on Days 1 - 28 plus azacitidine 75 mg/m2 SC or IV daily for 7 days. Cycle Length: 28 Days.

Subjects will continue treatment until subsequent alloSCT, documented morphological bone marrow and/or extramedullary disease progression, toxicity, withdrawal of consent, or the subject meets other protocol criteria for discontinuation (whichever occurs first).

After each cycle, MRD will be evaluated. AlloSCT is recommended at any time of MRD-negativity. After 6 cycles of treatment, regardless MRD status, patients will proceed to alloSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age
2. Subject must have received previous diagnosis of NPM1mut AML with or without concomitant FLT3-TKD or FLT3-ITD
3. At screening, subject must have confirmed NPM1 type A, B, or D mutant transcripts
4. Subject must be eligible for alloSCT, according to transplant center policy
5. Subject must have undergone at least two cycles of conventional anthracycline- and cytarabine-based chemotherapy, achieving first CR (CR1)
6. Subject must be in morphological CR1 with bone marrow detectable minimal residual disease (MRD) positivity, defined as qRT-PCR NPM1 transcript ≥ 0.01/100 ABL1 copies and confirmed in two consecutive determinations performed at 2 to 4 weeks' distance

   1. Molecular progression is defined in patients with molecular persistence at low copy number as an increase of MRD copy number ≥ 1 log10 between 2 positive samples.
   2. Molecular relapse is defined in patients previously tested MRD negative as an increase in MRD copy number ≥ 1 log10 between 2 positive samples
7. Subject must have a projected life expectancy of at least 12 weeks.
8. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status < 2
9. Subject must have adequate renal and hepatic function per local laboratory reference range as follows:

   * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0X ULN
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
   * Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours' urine collection.
10. Female subjects of childbearing potential must have negative results for pregnancy test at screening
11. Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from screening through 3 months after the end of treatment.
12. Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

1. Subject has acute promyelocytic leukemia (APL)
2. Subject has known active CNS involvement with AML
3. Subject has received previous treatment with venetoclax and/or hypomethylating agents
4. Subject has undergone alloSCT for AML
5. Subject has more than 5% of bone marrow blast cells at screening bone marrow aspirate
6. Subject is known to be positive for HIV
7. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
   2. Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
8. Cardiac history of CHF requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina;
9. DLCO ≤ 65% or FEV1 ≤ 65%;
10. Creatinine clearance < 30 ml/min
11. Subject has a cardiovascular disability status of New York Heart Association Class > 2

    a. Class 2 is i. defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity ii. results in fatigue, palpitations, dyspnea, or anginal pain
12. Patients who are pregnant or breast feeding and adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to administration of induction therapy). Post-menopausal women must be amenorrhoic for at least 12 months to be considered of non-child bearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drugs.
13. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy in terms of relapse rate | at 6 months
  Evaluation of treatment efficacy in terms of percentage of patients who do not experience overt relapse at 6 months or within stem cell transplant.

CONTACTS AND LOCATIONS:
Locations (1):
- EMATOLOGIA- AOU Policlinico S.Orsola, Bologna, Italy

REFERENCES:
- [Derived] Sartor C, Brunetti L, Audisio E, Cignetti A, Zannoni L, Cristiano G, Nanni J, Ciruolo R, Zingarelli F, Ottaviani E, Patuelli A, Bandini L, Forte D, Sciabolacci S, Cardinali V, Papayannidis C, Cavo M, Martelli MP, Curti A. A venetoclax and azacitidine bridge-to-transplant strategy for NPM1-mutated acute myeloid leukaemia in molecular failure. Br J Haematol. 2023 Aug;202(3):599-607. doi: 10.1111/bjh.18887. Epub 2023 May 24. PMID 37226312